CLINICAL TRIAL: NCT02941367
Title: International, Randomized, Open Label Study to Compare the Safety and Efficacy of Lixisenatide vs. Sulfonylurea on Top of Basal Insulin Treatment in Type 2 Diabetes Mellitus Subjects Who Elect to Fast During Ramadan
Brief Title: Safety Assessment of Lyxumia (Lixisenatide) and Sulfonylurea as Add-on Treatment to Basal Insulin in Uncontrolled Patients With Type 2 Diabetes Mellitus Who Elect to Fast During Ramadan
Acronym: LixiRam
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LPS14410; U1111-1172-3026 (Other: UTN)
Record Dates: First submitted 2016-10-12; First posted 2016-10-21 (Estimated); Last update posted 2022-04-25 (Actual); Status verified 2022-04

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — lixisenatide; Sulfonylurea Compounds; Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lyxumia (Experimental): Patients will receive Lyxumia once daily as investigational medicinal product (IMP) on top of patient's previous basal insulin with/without metformin. Non-IMPs will be administrated as per Investigator's indications according to local labeling, guidelines, and clinical judgment.
  Interventions: Drug: Lixisenatide (AVE0010); Drug: metformin; Drug: basal insulin
- Sulfonylurea (Active Comparator): Patients will continue the treatment with previous Sulfonylurea as IMP on top of patient's previous basal insulin with/without metformin. The IMP and non-IMPs will be administrated as per Investigator's indications according to local labeling, guidelines, and clinical judgment.
  Interventions: Drug: Sulfonylurea; Drug: metformin; Drug: basal insulin

INTERVENTIONS:
Drug: Lixisenatide (AVE0010) — Pharmaceutical form: solution for injection
  Route of administration: subcutaneous
  Other Names: Lyxumia
  Arms: Lyxumia
Drug: Sulfonylurea — Pharmaceutical form: tablet
  Route of administration: oral
  Arms: Sulfonylurea
Drug: metformin — Pharmaceutical form: tablet
  Route of administration: oral
Drug: basal insulin — Pharmaceutical form: solution for injection
  Route of administration: subcutaneous

SUMMARY:
Primary Objective:

To compare the safety, in terms of percentage of patients with symptomatic documented hypoglycemia during Ramadan fast, of lixisenatide versus sulfonylurea (SU).

Secondary Objectives:

* To assess effect of lixisenatide versus SU on:
* Changes in glycemic control;
* Changes in body weight.
* To assess overall safety of lixisenatide and SU.

DETAILED DESCRIPTION:
The total study duration per patient will have a minimum 12 weeks and maximum 22 weeks (up to 2 weeks screening period + 8-12 weeks pre-Ramadan period + 29-30 days Ramadan + 0 4 weeks post-Ramadan period). This is a phase 3b study in Kingdom of Saudi Arabia and Bangladesh (instead of phase 4 for other countries).

ELIGIBILITY:
Inclusion criteria :

* Patients with type 2 diabetes mellitus, diagnosed for at least 1 year at the time of the screening visit, insufficiently controlled with basal insulin + SU (≤50% max allowed dose) ±1 oral antidiabetic (OAD) drug.
* Patients who express the intention to fast during Ramadan.
* Signed informed consent.

Exclusion criteria:

* At the time of screening age < legal age of majority.
* Glycated hemoglobin (HbA1c) at screening visit: <7.5% or >10%.
* Body mass index (BMI) <20kg/m^2.
* Treatment with basal insulin for less than 6 months prior to screening.
* Prior antidiabetic medication (basal insulin and OADs) not at stable dose (eg, same medication, frequency and <20% dose change) in the last 8 weeks prior to screening.
* Previous treatment with short or rapid acting insulin other than for short term use (≤10 days) in relation to hospitalization or an acute illness in the last 6 months prior to screening.
* Any discontinuation from a glucagon like peptide-1 receptor agonist (GLP-1 RA) due to safety/tolerability issue or lack of efficacy.
* Patient not willing to perform self-monitored plasma glucose (SMPG) as required by protocol and to follow the instructions provided.
* Type 1, gestational or secondary diabetes.
* History of diabetic ketoacidosis.
* History of hypoglycemia unawareness.
* Any medical contraindication for sustained and safe fasting.
* Pregnant or breast-feeding women.
* Women of childbearing potential (WOCB) not protected by highly effective contraceptive method(s) of birth control and/or who are unwilling or unable to be tested for pregnancy.
* Known hypersensitivity/intolerance to lixisenatide (Lyxumia) or any of its excipients.
* All contraindications of the comparator and protocol mandated background therapies or warning/precaution of use (when appropriate) as displayed in the respective National Product Labeling.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 184 (Actual)
Dates: Start 2017-02-23 (Actual); Primary Completion 2017-08-04 (Actual); Study Completion 2017-08-04 (Actual)

PRIMARY OUTCOMES:
Percentage of patients with at least 1 documented symptomatic hypoglycemia event (plasma glucose ≤70 mg/dL; 3.9 mmol/L) | Approximately 30 days (from start to end of Ramadan holy month)

SECONDARY OUTCOMES:
Mean change in HbA1c | Baseline, 0-4 weeks pre- and 0-4 weeks post-Ramadan
Mean change in body weight | Baseline, 0-4 weeks pre- and 0-4 weeks post-Ramadan
Percentage of patients with 2-hour post prandial glucose (2hPPG) <180 mg/dL (10 mmol/L) | Last 14 days of Ramadan month
Percentage of patients with HbA1C <7% | At 0-4 weeks pre- and 0-4 weeks post-Ramadan
Percentage of patients with fasting plasma glucose (FPG) <130 mg/dL (7.22 mmol/L) | At pre-Ramadan visit
Percentage of patients with HbA1c <7%, no weight gain and no documented symptomatic hypoglycemia (plasma glucose ≤70 mg/dL; 3.9 mmol/L) | At 0-4 weeks pre- and 0-4 weeks post-Ramadan

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (16):
- India (12):
  - Investigational Site Number 356005, Ahmedabad
  - Investigational Site Number 356002, Bangalore
  - Investigational Site Number 356015, Bangalore
  - Investigational Site Number 356008, Bangalore
  - Investigational Site Number 356009, Hyderabad
  - Investigational Site Number 356018, Hyderabad
  - Investigational Site Number 356010, Hyderabad
  - Investigational Site Number 356003, Hyderabad
  - Investigational Site Number 356007, Jaipur
  - Investigational Site Number 356019, Madurai
  - Investigational Site Number 356014, Mumbai
  - Investigational Site Number 356022, Nagpur
- Israel (2):
  - Investigational Site Number 376001, Haifa
  - Investigational Site Number 376002, Safed
- Investigational Site Number 414001, Kuwait City, Kuwait
- Investigational Site Number 792002, Zonguldak, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- [Derived] Lee SWH, Chen WS, Sellappans R, Md Sharif SB, Metzendorf MI, Lai NM. Interventions for people with type 2 diabetes mellitus fasting during Ramadan. Cochrane Database Syst Rev. 2023 Jul 12;7(7):CD013178. doi: 10.1002/14651858.CD013178.pub2. PMID 37435938
- [Derived] Sahay R, Hafidh K, Djaballah K, Coudert M, Azar S, Shehadeh N, Hanif W, Hassanein M. Safety of lixisenatide plus basal insulin treatment regimen in Indian people with type 2 diabetes mellitus during Ramadan fast: A post hoc analysis of the LixiRam randomized trial. Diabetes Res Clin Pract. 2020 May;163:108148. doi: 10.1016/j.diabres.2020.108148. Epub 2020 Apr 14. PMID 32302665